CLINICAL TRIAL: NCT01135459
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of a 200-mcg Dose of CEP-33457 in Patients With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Efficacy and Safety of CEP-33457 in Participants With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C33457/2047
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — spliceosomal peptide P140

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CEP-33457 (Experimental): Participants will receive CEP-33457 200 mcg SC every 4 weeks for 20 weeks (Day 1, Weeks 4, 8, 12, 16, and 20).
  Interventions: Drug: CEP-33457
- Placebo (Placebo Comparator): Participants will receive placebo matching to CEP-33457 SC every 4 weeks for 20 weeks (Day 1, Weeks 4, 8, 12, 16, and 20).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CEP-33457 — CEP-33457 will be administered per dose and schedule specified in the arm description.
  Other Names: Lupuzor
  Arms: CEP-33457
Drug: Placebo — Placebo matching to CEP-33457 will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a 200 micrograms (mcg) dose of CEP-33457 compared with placebo in participants with active systemic lupus erythematosus (SLE) as assessed by the proportion of participants achieving a combined clinical response using the SLE responder index (SRI) at Week 24.

DETAILED DESCRIPTION:
The study consisted of a 2-week screening period (visit 1), a 20-week treatment period beginning with a baseline visit in which randomization was completed and study drug treatment began (visits 2 through 7), and a final assessment was performed 4 weeks after the last dose of study drug (visit 8 [week 24 or early termination]). Participants were randomized to receive either CEP-33457 or placebo subcutaneously (SC) every 4 weeks. Plasma samples for measurement of study drug concentration were collected in a subset of participants and study drug was administered at each study visit until the final visit. The dose of background steroid medication may have been increased, if needed, to treat the participant for minor fluctuations in lupus disease activity. One interim analysis was conducted when at least 80 participants completed Week 12 or had been withdrawn from the study. Participants who completed the treatment period returned to the study center 4 weeks after the last dose had been administered for final procedures and assessments. Final procedures and assessments for participants who withdrew from the study before 20 weeks of treatment were performed at the last visit. Final procedures and assessments for participants who participated in the study beyond week 24 were to be performed at the next regularly scheduled visit. Participants who complete the study will be eligible for participation in the 12-month open-label study (study C33457/3075; herein referred to as study 3075) to assess continued effectiveness and safety of the CEP-33457 treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participant has an established diagnosis of systemic lupus erythematosus (SLE) as defined by ACR Classification Revised Criteria. The diagnosis is fulfilled provided that at least 4 criteria are met.
* The participant has a positive test for antinuclear antibody (ANA) at screening and/or a positive test for anti-double-stranded deoxyribonucleic acid antibody (anti-dsDNA Ab) at screening.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, using a medically accepted method of contraception, and must agree to continued use of this method for the duration of the study and for 30 days after discontinuation of study drug treatment.
* The participant has a clinical SLEDAI-2K score of at least 6 points during screening.
* The participant does not have an "A" score on the BILAG-2004 scale.
* If the patient is using oral corticosteroids, the weekly cumulative dose must not exceed 80 mg of prednisone equivalent; the weekly dose must be stable over the 4 weeks preceding the first dose of study drug.
* If the participant is using antimalarials, methotrexate, leflunomide, mycophenolate mofetil, or azathioprine, the start date must be at least 3 months prior to the first dose of study drug, and the daily dose must be stable over the 4 weeks preceding the first dose of study drug.
* If the participant is not currently using corticosteroids, antimalarials, methotrexate, mycophenolate mofetil, or azathioprine, the last dose (in case of previous use) must be at least 4 weeks prior to the first dose of study drug. For leflunomide, the stop date must be at least 8 weeks before the first dose of study drug, unless an adequate cholestyramine washout has been completed.

Exclusion Criteria:

* The participant has been treated with intramuscular or intravenous (iv) pulse steroids (ie, 250 to 1000 milligrams [mg] iv total daily dose of methylprednisolone) within 4 weeks of the first dose of study drug. The use of intra-articular steroids may be allowed after consultation with the medical expert.
* The participant has received tacrolimus, cyclosporine A, or iv immunoglobulins (IVIG) within 3 months of the first dose of study drug.
* The participant has received cyclophosphamide within 12 months prior to the first dose of study drug.
* The participant has been treated for SLE with agents such as fusion proteins, therapeutic proteins, or monoclonal antibodies or antibody fragments, within 12 months of the first dose of study drug.
* The participant has received B-cell depleting agents such as rituximab and has not yet normalized the B-cell count (ie, CD20+ B-cell count is less than 200 and the absolute lymphocyte count [ALC] is less than 1500/μL).
* The participant has New York Heart Association (NYHA) Class III or IV congestive heart failure.
* The participant has severe active lupus nephritis or cerebritis.
* The participant has an estimated glomerular filtration rate (eGFR) of less than 30 milliliters (mL)/minute (min)/1.73 square meter (m^2) (via Modification of Diet in Renal Disease [MDRD] equation).
* The participant has an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value greater than 2 times the upper limit of normal (ULN) or a total bilirubin level greater than 1.5 times ULN.
* The participant has a planned immunization with a live or live attenuated vaccine within 3 months prior to administration of the first dose of study drug and for 3 months after administration of the last dose of study drug.
* The participant has any clinically significant abnormalities on electrocardiogram (ECG) that are not related to SLE, as determined by the investigator. Participant with stable ECG changes without evidence of active cardiovascular disease may participate at the discretion of the investigator and medical monitor.
* The participant has an ongoing active systemic infection requiring treatment or a history of severe infection, such as hepatitis or pneumonia, in the 3 months prior to administration of the first dose of study drug. Less severe infections in the 3 months prior to administration of the first dose of study drug are permitted at the discretion of the investigator and medical monitor.
* The participant has any concomitant medical condition unrelated to SLE that may interfere with his or her safety or with evaluation of the study drug, as determined by the investigator.
* The participant has a history of a medical condition other than SLE that has required treatment with steroids in excess of 80 mg of prednisone equivalent/week within 6 months of the first dose of study drug.
* The participant has a positive test result for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C (HCV Ab).
* The participant has a known positive history of antibodies to human immunodeficiency virus (HIV) or HIV disease.
* The participant has a history of alcohol or substance dependence or abuse (with the exception of nicotine), according to the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, Fourth Edition, Text Revision (DSM-IV-TR), within 3 months of the screening visit or has current substance abuse.
* The participant has a history of severe allergic reactions to or hypersensitivity to any component of the study drug or placebo.
* The participant has undergone or is undergoing treatment with another investigational drug for the treatment of lupus within 6 months prior to the 1st dose of study drug or has received any other investigational drug for any other condition within 30 days prior to the 1st dose of study drug.
* The participant has previously participated in a Cephalon- or ImmuPharma-sponsored clinical study with CEP-33457.
* The participant is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The participant is unlikely to comply with the study protocol or is unsuitable for any other reason, as judged by the investigator or medical monitor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-06-24 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2012-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (86):
- United States (40):
  - Teva Investigational Site 27, Birmingham, Alabama
  - Teva Investigational Site 20, Tucson, Arizona
  - Teva Investigational Site 16, Los Angeles, California
  - Teva Investigational Site 5, Los Angeles, California
  - Teva Investigational Site 7, San Diego, California
  - Teva Investigational Site 14, San Leandro, California
  - Teva Investigational Site 17, Stanford, California
  - Teva Investigational Site 30, Aurora, Colorado
  - Teva Investigational Site 4, Aventura, Florida
  - Teva Investigational Site 32, Clearwater, Florida
  - Teva Investigational Site 35, Fort Lauderdale, Florida
  - Teva Investigational Site 1, Jupiter, Florida
  - Teva Investigational Site 11, Tampa, Florida
  - Teva Investigational Site 8, Atlanta, Georgia
  - Teva Investigational Site 31, Atlanta, Georgia
  - Teva Investigational Site 38, Stockbridge, Georgia
  - Teva Investigational Site 23, Coeur d'Alene, Idaho
  - Teva Investigational Site 37, Lexington, Kentucky
  - Teva Investigational Site 36, Baltimore, Maryland
  - Teva Investigational Site 10, Boston, Massachusetts
  - Teva Investigational Site 22, Ann Arbor, Michigan
  - Teva Investigational Site 9, Manhasset, New York
  - Teva Investigational Site 3, Chapel Hill, North Carolina
  - Teva Investigational Site 28, Charlotte, North Carolina
  - Teva Investigational Site 18, Durham, North Carolina
  - Teva Investigational Site 2, Monroe, North Carolina
  - Teva Investigational Site 21, Oklahoma City, Oklahoma
  - Teva Investigational Site 13, Oklahoma City, Oklahoma
  - Teva Investigational Site 25, Duncansville, Pennsylvania
  - Teva Investigational Site 26, Pittsburgh, Pennsylvania
  - Teva Investigational Site 15, Charleston, South Carolina
  - Teva Investigational Site 29, Dallas, Texas
  - Teva Investigational Site 40, Houston, Texas
  - Teva Investigational Site 6, Houston, Texas
  - Teva Investigational Site 39, Mesquite, Texas
  - Teva Investigational Site 34, San Antonio, Texas
  - Teva Investigational Site 24, Temple, Texas
  - Teva Investigational Site 19, Arlington, Virginia
  - Teva Investigational Site 12, Seattle, Washington
  - Teva Investigational Site 33, Milwaukee, Wisconsin
- Belgium (3):
  - Teva Investigational Site 102, Brussels
  - Teva Investigational Site 101, Liège
  - Teva Investigational Site 100, Yvoir
- Czechia (4):
  - Teva Investigational Site 201, Brno
  - Teva Investigational Site 200, Olomouc
  - Teva Investigational Site 202, Prague
  - Teva Investigational Site 203, Prague
- France (5):
  - Teva Investigational Site 301, Lille
  - Teva Investigational Site 302, Nantes
  - Teva Investigational Site 300, Paris
  - Teva Investigational Site 303, Paris
  - Teva Investigational Site 304, Strasbourg
- Germany (7):
  - Teva Investigational Site 402, Aachen
  - Teva Investigational Site 403, Berlin
  - Teva Investigational Site 401, Dresden
  - Teva Investigational Site 404, Düsseldorf
  - Teva Investigational Site 406, Hamburg
  - Teva Investigational Site 405, Mainz
  - Teva Investigational Site 400, München
- Hungary (3):
  - Teva Investigational Site 501, Budapest
  - Teva Investigational Site 502, Debrecen
  - Teva Investigational Site 500, Zalaegerszeg
- Poland (7):
  - Teva Investigational Site 603, Dąbrówka
  - Teva Investigational Site 600, Elblag
  - Teva Investigational Site 602, Gmina Końskie
  - Teva Investigational Site 604, Lublin
  - Teva Investigational Site 601, Lublin
  - Teva Investigational Site 606, Warsaw
  - Teva Investigational Site 605, Wroclaw
- Portugal (4):
  - Teva Investigational Site 701, Amadora
  - Teva Investigational Site 702, Coimbra
  - Teva Investigational Site 703, Porto
  - Teva Investigational Site 700, Porto
- Spain (3):
  - Teva Investigational Site 751, Dresden
  - Teva Investigational Site 752, Santander
  - Teva Investigational Site 750, Seville
- Ukraine (6):
  - Teva Investigational Site 901, Donetsk
  - Teva Investigational Site 905, Ivano-Frankivsk
  - Teva Investigational Site 900, Kyiv
  - Teva Investigational Site 902, Kyiv
  - Teva Investigational Site 903, Kyiv
  - Teva Investigational Site 904, Lviv
- United Kingdom (4):
  - Teva Investigational Site 803, Bath
  - Teva Investigational Site 801, Leeds
  - Teva Investigational Site 800, London
  - Teva Investigational Site 802, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to CEP-33457 subcutaneously (SC) every 4 weeks for 20 weeks (Day 1, Weeks 4, 8, 12, 16, and 20).
- CEP-33457: Participants received CEP-33457 200 micrograms (mcg) SC every 4 weeks for 20 weeks (Day 1, Weeks 4, 8, 12, 16, and 20).
Period: Overall Study
Arm/Group | Placebo | CEP-33457
Started | 92 | 91
Received at Least 1 Dose of Study Drug | 92 | 91
Completed | 71 | 71
Not Completed | 21 | 20
Not completed — Adverse Event | 8 | 10
Not completed — Lack of Efficacy | 3 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 5 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Non-compliance to study procedures | 0 | 1
Not completed — Other than specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received placebo matched to CEP-33457 SC every 4 weeks for 20 weeks (Day 1, Weeks 4, 8, 12, 16, and 20).
- CEP-33457: Participants received CEP-33457 200 mcg SC every 4 weeks for 20 weeks (Day 1, Weeks 4, 8, 12, 16, and 20).
- Total: Total of all reporting groups
Arm/Group | Placebo | CEP-33457 | Total
Number analyzed (Participants) | 92 | 91 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.88) | 42.0 (11.25) | 41.0 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 86 | 169
  Male | 9 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 82 | 80 | 162
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 64 | 67 | 131
  Race: Black | 17 | 18 | 35
  Race: Asian | 3 | 2 | 5
  Race: American Indian or Alaskan Native | 0 | 1 | 1
  Race: Other | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Combined Clinical Response Using the Systemic Lupus Erythematosus (SLE) Responder Index (SRI) at Week 24
Description: An SRI response was defined as a reduction from baseline in SLE Disease Activity Index 2000 (SLEDAI-2K) score of ≥4 points, no worsening in Physician Global Assessment (PhGA), no new British Isles Lupus Assessment Group (BILAG) A body system score, and ≤1 new BILAG B body system score from baseline. SLEDAI-2K includes 24 weighted clinical and laboratory variables. Total score = 0 to 105. A score of 6 to 10 = moderate disease activity, and a reduction of >3 points = improvement. PhGA was completed by physician using a visual analog scale (VAS) from 0=none to 3=severe. A change of >0.3 points = worsening. BILAG includes 97 clinical and laboratory items. Each organ system is assigned a score displayed as a grade from A to E: A=very active disease; B=patient needs increase in treatment for moderately active disease; C=stable or mild disease; D=previous organ involvement but no current disease activity; and E=no current disease activity and organ system has never been involved.
Time Frame: Week 24
Population: Full analysis set included all randomized participants who took at least 1 dose of study drug and had the baseline SLEDAI-2K total score, BILAG 2004 body system scores, and the PhGA score.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
Participants | 37 | 31
Statistical Analysis 1: Comparison: Placebo vs CEP-33457; Analysis was performed using a logistic regression model with treatment and stratification factors as main factors; Test type: Other; p = 0.3989, Regression, Logistic; Odds Ratio (OR) = 0.7649, 95% CI 2-sided [0.4 to 1.4]

2. Secondary Outcome: Number of Participants Achieving an SRI Response at Each Visit During the Treatment Period
Description: An SRI response was defined as a reduction from baseline in SLEDAI-2K score of ≥4 points, no worsening in PhGA, no new BILAG A body system score, and ≤1 new BILAG B body system score from baseline. SLEDAI-2K includes 24 weighted clinical and laboratory variables. Total score = 0 to 105. A score of 6 to 10 = moderate disease activity, and a reduction of >3 points = improvement. PhGA was completed by physician using a VAS from 0=none to 3=severe. A change of >0.3 points = worsening. BILAG includes 97 clinical and laboratory items. Each organ system is assigned a score displayed as a grade from A to E: A=very active disease; B=participant needs increase in treatment for moderately active disease; C=stable or mild disease; D=previous organ involvement but no current disease activity; and E=no current disease activity and organ system has never been involved.
Time Frame: Weeks 4, 8, 12, 16, and 20
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
Participants
  Week 4 | 11 | 13
  Week 8 | 19 | 27
  Week 12 | 33 | 29
  Week 16 | 29 | 28
  Week 20 | 38 | 30

3. Secondary Outcome: Number of Participants Achieving a Reduction of at Least 4 Points in the SLEDAI-2K Total Score
Description: The SLEDAI-2K is a global index and includes 24 weighted clinical and laboratory variables. The total score (sum of all 24 scores) ranges from 0 to 105. A SLEDAI-2K score of 6 to 10 is indicative of moderate disease activity, and improvement is defined as a reduction of more than 3 points.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
Participants | 40 | 32

4. Secondary Outcome: Number of Participants Achieving a British Isles Lupus Assessment Group (BILAG) 2004 Response
Description: The BILAG 2004 is a validated objective and subjective global measure of the disease activity of SLE based on the physician intention to treat. It includes 97 clinical and laboratory items to evaluate SLE disease activity in 9 organ systems; each organ system is assigned a score displayed as a grade from A to E, as follows: A=very active disease; B=participant needs increase in treatment for moderately active disease; C=stable or mild disease; D=previous organ involvement but no current disease activity; and E=no current disease activity and the organ system has never been involved. BILAG 2004 response was defined as no new A body system score and no more than 1 new BILAG B body system score from baseline.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
Participants
  Week 4 | 86 | 82
  Week 8 | 82 | 79
  Week 12 | 80 | 75
  Week 16 | 76 | 66
  Week 20 | 74 | 66
  Week 24 | 70 | 63

5. Secondary Outcome: Number of Participants Achieving a BILAG 2004 Clinical Response
Description: The BILAG 2004 is a validated objective and subjective global measure of the disease activity of SLE based on the physician intention to treat. It includes 97 clinical and laboratory items to evaluate SLE disease activity in 9 organ systems; each organ system is assigned a score displayed as a grade from A to E, as follows: A=very active disease; B=participant needs increase in treatment for moderately active disease; C=stable or mild disease; D=previous organ involvement but no current disease activity; and E=no current disease activity and the organ system has never been involved. BILAG 2004 clinical response was defined as having an improvement in at least 1 category from a B score at baseline to a C or D score with no worsening in any other category from baseline.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
Participants
  Week 4 | 32 | 36
  Week 8 | 34 | 37
  Week 12 | 45 | 34
  Week 16 | 42 | 33
  Week 20 | 43 | 32
  Week 24 | 39 | 31

6. Secondary Outcome: Number of Participants Achieving a Physician Global Assessment (PhGA) Response
Description: The PhGA was completed by the physician using a 3 inch VAS labeled from 0=none to 3=severe. The PhGA response was defined as having no worsening in PhGA (with worsening defined as an increase in PhGA of more than 0.30 inch from baseline).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
Participants
  Week 4 | 80 | 76
  Week 8 | 83 | 75
  Week 12 | 77 | 68
  Week 16 | 71 | 61
  Week 20 | 73 | 64
  Week 24 | 71 | 67

7. Secondary Outcome: Number of Participants Achieving a Patient's Global Assessment (PtGA) Response
Description: The PhGA was completed by the participant using a 3 inch VAS labeled from 0=none to 3=severe. The PtGA response was defined as having no worsening in PtGA (with worsening defined as an increase in PtGA of more than 0.30 inch from baseline).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
Participants
  Week 4 | 79 | 65
  Week 8 | 73 | 67
  Week 12 | 64 | 63
  Week 16 | 65 | 57
  Week 20 | 65 | 59
  Week 24 | 63 | 59

8. Secondary Outcome: Change From Baseline in the Medical Outcome Survey Short-Form 36 (SF-36) Patient-Reported Questionnaire For Physical Component Summary (PCS) Score at Weeks 12 and 24
Description: The SF-36 questionnaire has 36 questions composing the scale that represent 8 domains: 1) physical functioning, role physical, 2) bodily pain, 3) general health, 4) vitality, 5) social functioning, 6) role, 7) emotional, and 8) mental health. The scores for the 8 domains were combined into two summary scores: the physical component summary (PCS) score and the mental component summary (MCS) score. Items 1 to 4 primarily contribute to the PCS score of the SF-36. Items 5-8 primarily contribute to the MCS score of the SF-36. Scores on each item were summed and averaged (range: 0=worst to 100=best). Higher scores represent better health status and functional ability.
Time Frame: Baseline, Week 12, Week 24
Population: Full analysis set included all randomized participants who took at least 1 dose of study drug and had the baseline SLEDAI-2K total score, BILAG 2004 body system scores, and the PhGA score. Overall number of participants analyzed = participants evaluable for this outcome measure. Number analyzed = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 89
units on a scale
  Baseline | 37.3 (9.60) | 36.1 (10.06)
  Change at Week 12: number analyzed (Participants) | 82 | 78
  Change at Week 12 | 2.5 (6.69) | 2.2 (6.70)
  Change at Week 24: number analyzed (Participants) | 72 | 70
  Change at Week 24 | 2.1 (7.66) | 2.4 (8.36)

9. Secondary Outcome: Change From Baseline in the Medical Outcome Survey SF-36 Patient-Reported Questionnaire For Mental Component Summary (MCS) Score at Weeks 12 and 24
Description: as for outcome 8
Time Frame: Baseline, Week 12, Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 89
units on a scale
  Baseline | 40.6 (12.99) | 41.7 (12.26)
  Change at Week 12: number analyzed (Participants) | 82 | 78
  Change at Week 12 | 0.5 (11.10) | 1.0 (9.66)
  Change at Week 24: number analyzed (Participants) | 72 | 70
  Change at Week 24 | 0.4 (10.45) | 1.7 (10.81)

10. Secondary Outcome: Systemic Lupus International Collaborative Clinics/American College of Rheumatology (SLICC/ACR) Damage Index
Description: SLICC/ACR score or damage index is a measure of cumulative damage due to SLE. Damage is defined as nonreversible change (not related to active inflammation) occurring since onset of lupus, ascertained by clinical assessment and present for at least 6 months. Damage is defined for 12 separate organ systems: ocular (range 0-2), neuropsychiatric (0-6), renal (0-3), pulmonary (0-5), cardiovascular (0-6), peripheral vascular (0-5), gastrointestinal (0-6), musculoskeletal (0-7), skin (0-3), endocrine (diabetes) (0-1), gonadal (0-1) and malignancies (0-2). A score of 0=no damage, early damage is defined as ≥1. The total maximum score is 47, and increasing score indicates increasing disease damage severity.
Time Frame: Baseline, Week 24
Population: Full analysis set included all randomized participants who took at least 1 dose of study drug and had the baseline SLEDAI-2K total score, BILAG 2004 body system scores, and the PhGA score. Number analyzed = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 90
units on a scale
  Baseline | 0.7 (1.30) | 0.6 (1.08)
  Change at Week 24: number analyzed (Participants) | 74 | 70
  Change at Week 24 | -0.1 (0.47) | -0.1 (0.37)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 24
Population: Safety analysis set included all randomized participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CEP-33457
Number analyzed (Participants) | 92 | 91
Participants | 81 | 77

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: Safety analysis set included all randomized participants who took at least 1 dose of study drug.
Arm/Group | Placebo | CEP-33457
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/91
Serious Adverse Events (participants affected / at risk) | 13/92 | 9/91
Other Adverse Events (participants affected / at risk) | 58/92 | 61/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | CEP-33457 (N=91)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | CEP-33457 (N=91)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 6 (10)
Nausea (Gastrointestinal disorders) | 7 (11) | 5 (7)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (7)
Fatigue (General disorders) | 4 (5) | 6 (7)
Injection site erythema (General disorders) | 1 (1) | 7 (23)
Pyrexia (General disorders) | 7 (10) | 4 (5)
Nasopharyngitis (Infections and infestations) | 7 (7) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 7 (9)
Urinary tract infection (Infections and infestations) | 9 (10) | 3 (6)
Contusion (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Weight decreased (Investigations) | 5 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 12 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (9) | 16 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 9 (16) | 11 (14)
Headache (Nervous system disorders) | 9 (9) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 12 (22) | 11 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.